CLINICAL TRIAL: NCT02292979
Title: Brentuximab Vedotin Associated With Chemotherapy in Untreated Patients With Stage I/II Unfavourable Hodgkin Lymphoma. A Randomized Phase II LYSA-FIL-EORTC Intergroup Study
Brief Title: Brentuximab Vedotin Associated With Chemotherapy in Untreated Patients With Hodgkin Lymphoma.
Acronym: BREACH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREACH
Record Dates: First submitted 2014-10-28; First posted 2014-11-18 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Hodgkin Lymphoma
Keywords: HL
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABVD (Active Comparator): Patients in standard arm receive Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine on Day 1 and D14 of each 4-week-cycle during 4 cycles
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine
- AVD+BV (Experimental): Patients in experimental arm receive Doxorubicin, Vinblastine, Dacarbazine and Brentuximab vedotin on Day 1 and D14 of each 4-week-cycle during 4 cycles
  Interventions: Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Doxorubicin — 25mg/m2
Drug: Bleomycin — 10mg/m2
  Arms: ABVD
Drug: Vinblastine — 6mg/m2
Drug: Dacarbazine — 375mg/m2
Drug: Brentuximab Vedotin — 1.2 mg/kg
  Arms: AVD+BV

SUMMARY:
This study aims to evaluate the efficacy of brentuximab vedotin + AVD combination (doxorubicine, vinblastine, dacarbazine) in patients with Hodgkin lymphoma stage I / II with an unfavorable diagnosis, assessed by the negativity of PET (positron emission tomography ) after two cycles of chemotherapy.

DETAILED DESCRIPTION:
Patients will receive either ABVD chemotherapy (standard treatment = doxorubicin, bleomycin, vinblastine, dacarbazine) or the Brentuximab vedotin in combination with chemotherapy AVD (study treatment), depending on randomization. Radiotherapy is planned after chemotherapy or immunochemotherapy.

PET scans will be performed before inclusion, after 2 cycles of chemotherapy and after 4 cycles of chemotherapy (if PET after two cycles was positive), at the end of treatment and during follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD30+ classical Hodgkin lymphoma
* Supradiaphragmatic Ann Arbor clinical stage I or II
* Previously untreated
* PET scan without IV contrast at diagnosis available for central review with at least one hypermetabolic lesion
* Unfavourable (U) characteristics according to the classic EORTC/LYSA clinical prognostic factors, including patients with at least one of the following factors:

  * CSII ≥ 4 nodal areas
  * age ≥ 50 yrs
  * M/T ratio ≥ 0.35
  * ESR ≥ 50 (without B-symptoms) or ESR ≥ 30 with B-symptoms
* ECOG performance status 0-2
* Life expectancy > 6 months
* Age 18 to 60 years
* Availability for periodic blood sampling, study-related assessments, and management of toxicity at the treating institution.
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, through 6 months after the last dose of study drug, OR agree to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized (ie, status postvasectomy), who:

  o Agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
* Written informed consent.
* Required baseline laboratory data:

  * Absolute neutrophil count ≥ 1,500/µL
  * Platelet count ≥ 75,000/ µL
  * Hemoglobin ≥ 8g/dL
  * Serum total bilirubin ≤ 1.5 X ULN unless the elevation is known to be due to Gilbert syndrome.
  * Serum creatinine ≤ 2.0 mg/dL and/or calculated creatinine clearance > 40 mL/minute (Cockcroft-Gault formula or MDRD)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 X ULN

Exclusion Criteria:

* Histological diagnosis different from classical Hodgkin Lymphoma. Nodular lymphocyte predominant subtypes (nodular paragranuloma or Poppema paragranuloma) are excluded.
* Known cerebral or meningeal disease of any etiology, including signs or symptoms of PML
* Any sensory or motor peripheral neuropathy ≥ Grade 2
* Known history of any of the following cardiovascular conditions

  * Myocardial infarction within 2 years of randomization
  * New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 14)
  * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Recent evidence (within 30 days before first dose of study drug) of a left-ventricular ejection fraction <50%
* Unstable diabetes mellitus (to avoid uninterpretable FDG-PET scan).
* Known HIV positive
* HCV positive
* HBV positive. This means:

  * HBsAg positive
  * HBsAg negative, anti-HBs positive and/or anti-HBc positive and detectable viral DNA (HBsAg negative patients and viral DNA negative and patients seropositive due to a history of hepatitis B vaccine are eligible).
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors. Carcinoma in situ of any type not excluded if complete resection.
* Dementia or altered mental status
* Pregnancy or breastfeeding.
* Previous treatment with any anti-CD30 antibody.
* Known hypersensitivity to any excipients contained in the BV formulation or known contra-indication to any drug contained in the chemotherapy regimens
* Treatment with corticosteroids before baseline PET scan
* Known active viral, bacterial, or fungal infection requiring treatment with antimicrobial therapy or with untreated known active Grade 3 viral, bacterial, or fungal infection, within 2 weeks prior to the first dose of BV
* Treatment with any investigational drug within 30 days before first cycle of treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
PET2 assessment | 8 weeks
  Assessment of PET after two cycles according to the five-point scale Deauville criteria (Negative = 1, 2, 3 and Positive = 4, 5), based on central review.

SECONDARY OUTCOMES:
Complete response (CR) rate | 16 weeks
  according to Cheson 2007 criteria
Progression free survival (PFS) | 5 years
  Survival without disease progression
Overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc André, Pr, Principal Investigator — Lymphoma Study Association; Luc Fornecker, Dr, Principal Investigator — Lymphoma Study Association
Locations (65):
- Belgium (11):
  - ZNA Middelheim, Antwerp
  - ZNA Stuivenberg, Antwerp
  - A.Z. Sint Jan AV, Bruges
  - Institut Jules Bordet, Brussels
  - UCL Louvain Saint Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - CHU de Liege, Liège
  - AZ Delta - Campus H. Hartziekenhuis, Roeselare
  - CHU Dinant Godinne, Yvoir
- University Hospital Rebro, Zagreb, Croatia
- Rigshospitalet, Copenhagen, Denmark
- France (43):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH de Annecy, Annecy
  - CHU Jean Minjoz, Besançon
  - CH de Bourg en Bresse, Bourg-en-Bresse
  - Centre François Baclesse, Caen
  - CHU de Caen, Caen
  - CH de Chalon sur Saône, Chalon-sur-Saône
  - CH de Chambéry, Chambéry
  - Hôpital Antoine Béclère, Clamart
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH Sud Francilien de Corbeil, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CH La Rochelle, La Rochelle
  - Centre Hospitalier de Versailles - André Mignot, Le Chesnay
  - CHRU de Lille - Hôpital Claude Hurriez, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CH de Meaux, Meaux
  - CHR de Metz, Metz
  - CHU de Montpellier - Saint Eloi, Montpellier
  - CHU de Mulhouse, Mulhouse
  - CHU Nancy Brabois, Nancy
  - CHU Hôtel Dieu Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - Hôpital Necker, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Centre François Magendie, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - CH de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Netherlands (9):
  - Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam
  - Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Reinier De Graaf Gasthuis, Delft
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Radboud University Medical Center Nijmegen, Nijmegen
  - Erasmus MC Cancer Institute - location Daniel den Hoed, Rotterdam
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldkuhle M, Kreuzberger N, von Tresckow B, Eichenauer DA, Specht L, Monsef I, Skoetz N. Chemotherapy alone versus chemotherapy plus radiotherapy for adults with early-stage Hodgkin's lymphoma. Cochrane Database Syst Rev. 2024 Dec 2;12(12):CD007110. doi: 10.1002/14651858.CD007110.pub4. PMID 39620432
- [Derived] Fornecker LM, Lazarovici J, Aurer I, Casasnovas RO, Gac AC, Bonnet C, Bouabdallah K, Feugier P, Specht L, Molina L, Touati M, Borel C, Stamatoullas A, Nicolas-Virelizier E, Pascal L, Lugtenburg P, Di Renzo N, Vander Borght T, Traverse-Glehen A, Dartigues P, Hutchings M, Versari A, Meignan M, Federico M, Andre M; LYSA-FIL-EORTC Intergroup. Brentuximab Vedotin Plus AVD for First-Line Treatment of Early-Stage Unfavorable Hodgkin Lymphoma (BREACH): A Multicenter, Open-Label, Randomized, Phase II Trial. J Clin Oncol. 2023 Jan 10;41(2):327-335. doi: 10.1200/JCO.21.01281. Epub 2022 Jul 22. PMID 35867960